CLINICAL TRIAL: NCT05094947
Title: Indwelling Urinary Catheterization Versus Clean Intermittent Catheterization for the Management of Acute Urinary Retention: Multicenter, Randomized, Controlled Clinical Trial.
Brief Title: Intermittent Catheterization Versus Trial Without Catheter
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Moscow State University of Medicine and Dentistry (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Moscow MSUMD
Record Dates: First submitted 2021-08-10; First posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-08

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Benign prostatic hyperplasia; acute urinary retention; intermittent catheterization; urethral catheter; trial without catheter
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Intermittent Urethral Catheterization; Clinical Trials as Topic; Catheters; Adrenergic alpha-Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intermittent catheterization (group B) (Experimental): Procedure/Surgery: The acute urinary retention in group B is managed by clean intermittent catheterization along with alpha-blockers during 3 period. After 3 days the ability of spontaneous voiding is assessed and registered as an outcome.
  Interventions: Procedure: intermittent catheterization; Drug: alpha-blockers
- Catheter Foley (group A) (Active Comparator): The acute urinary retention in group A is managed by trial without catheter along with alpha-blockers during 3 period. After 3 days the indwelling Foley catheter is removed and ability of spontaneous voiding is assessed and registered as an outcome.
  Interventions: Procedure: trial without catheter; Drug: alpha-blockers

INTERVENTIONS:
Procedure: intermittent catheterization — clean intermittent catheterization with catheter Nelaton
  Arms: intermittent catheterization (group B)
Procedure: trial without catheter — catheter Foley
  Arms: Catheter Foley (group A)
Drug: alpha-blockers — tamsulosin, alfuzosin, doxazosin, silodosin

SUMMARY:
This is a prospective, comparative, multicenter, randomized controlled trial. The aim of this study is to compare the efficacy, safety and quality of life within patients with acute urinary retention managed by the intermittent catheterization compared or indwelling Foley catheter.

ELIGIBILITY:
Inclusion Criteria:

Men with acute urinary retention due to prostatic hyperplasia

Exclusion Criteria:

* Patient's with serious conditions and incapacity
* Previous urethral or prostate surgery.
* Urethral stricture.
* Urethrorrhagia.
* Injuries of urethra and perineum.
* Attempts of bladder catheterization within 15 days before the acute urinary retention episode.
* Urinary tract infection.
* Neurogenic bladder.
* Chronic urinary retention with a bladder volume of more than 1 liter.
* Obstructive uropathy due to the acute urinary retention.

Ages: 21 Years to 95 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-08-03 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Assessment of the quality of life | 2 months
  Assessment of the quality of life according to the SF-36 questionnaire on the first, second, or third day after the start of intermittent catheterization

SECONDARY OUTCOMES:
Assessment of the restoration of self-urination. | 2 months
  A positive outcome is considered to be the restoration of independent urination, and the presence of no more than 150 ml of residual urine in a control study 12-24 hours after the restoration of urination.

CONTACTS AND LOCATIONS:
Overall Officials: Vigen Malkhasyan, Principal Investigator — Moscow state university of medicine and dentistry named after A.I. Evdokimov
Locations (1):
- Moscow state university of medicine and dentistry named after A.I. Evdokimov, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No